CLINICAL TRIAL: NCT02589223
Title: A Pilot Randomized Controlled Trial to Determine the Feasibility and Effectiveness of Early Multisensory Stimulation Intervention in Patients in the Trauma-Neurosurgical Intensive Care Unit (TNICU) Following Severe Acquired Brain Injury
Brief Title: A Trial to Determine the Feasibility and Effectiveness of Early Multisensory Stimulation Intervention in Patients in the Trauma-Neurosurgical Intensive Care Unit (TNICU) Following Severe Acquired Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Our enrollment numbers were low - very few eligible study subjects.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSS2015
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Traumatic Brain Injury With Prolonged Loss of Consciousness
Keywords: multisensory stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory Stimulation Group (Active Comparator): Intervention sessions will occur 3 times per week, for approximately 30 minutes per session for a total of 4 weeks. Subjects assigned to the multisensory stimulation group will receive the multisensory stimulation protocol designed for the study, which will include a variety of techniques designed to awaken the individual. Stimulus provided may include: visual activities (i.e. presenting the individual with objects/pictures to look at), auditory information (i.e. playing music or speaking), tactile stimuli (i.e. touching the individual with materials of different textures), taste and smell stimuli (i.e. offering items for the individual to taste or smell).
  Interventions: Other: Multisensory Stimulation
- Control Group (Placebo Comparator): Intervention sessions will occur 3 times per week, for approximately 30 minutes per session for a total of 4 weeks. During each session, subjects will be played a pre-recorded reading of complex material for 30 minutes, in order to assist with control/blinding.
  Interventions: Other: Control

INTERVENTIONS:
Other: Multisensory Stimulation — Subjects assigned to the multisensory stimulation group will receive the multisensory stimulation protocol designed for the study, which will include a variety of techniques designed to awaken the individual. Stimulus provided may include: visual activities (i.e. presenting the individual with objects/pictures to look at), auditory information (i.e. playing music or speaking), tactile stimuli (i.e. touching the individual with materials of different textures), taste and smell stimuli (i.e. offering items for the individual to taste or smell).
  Arms: Multisensory Stimulation Group
Other: Control — Intervention sessions will occur 3 times per week, for approximately 30 minutes per session for a total of 4 weeks. During each session, subjects will be played a pre-recorded reading of complex material for 30 minutes, in order to assist with control/blinding.
  Arms: Control Group

SUMMARY:
St. Michael's Hospital (SMH) provides service to individuals with some of the most severe brain injuries and intensive care needs in Canada. These patients often require prolonged intensive care admissions, lengthy hospital stays, involvement of many health professionals, and long-term support for ongoing care requirements. Many hospitals face resource limitations, specifically involving the health disciplines and their ability to provide frequent intervention.

It has been proposed that multisensory stimulation (i.e. exposing the patient to various sights, sounds, smells, etc.) in the early stages of brain injury recovery may result in improved responsiveness/cognitive function.

Previous research has indicated a potential benefit for early multisensory stimulation intervention for patients with severe brain injury. However there is still not enough conclusive evidence to confirm whether the intervention is truly effective. The investigators are proposing a pilot randomized controlled study (placebo-controlled, double-blinded) to determine the feasibility and examine the effectiveness of early multisensory stimulation with patients following severe brain injury who remain in a coma, vegetative state, or minimally conscious state. Eligible patients will be randomized to a control group (standard care + family/caregiver education) or an intervention group (standard care + family/caregiver education + early sensory intervention). Data regarding number of patients enrolled, amount of intervention completed, percentage of outcome data collected, patient's level of responsiveness and cognitive function will be collected before and after the intervention period, using several outcome measures. The investigators hope to determine the feasibility of conducting this type of study within this clinical setting and the effectiveness of multisensory stimulation with this patient population.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 weeks post injury, no more than 8 weeks post injury
* Glasgow Coma Scale score of less than or equal to 9, or motor component score of 5 or less if patient intubated
* No previous brain injury
* No chronic/progressive neurological illness
* No intracranial pressure monitor
* No more than1 pre-existing sensory impairment (e.g. deafness, blindness)
* Functional level of English for patient and Substitute Decision Maker (i.e. conversational English, work/education in English, completion of English as a Second Language course, etc.)
* Deemed medically appropriate as per Nurse Practitioner/MD (e.g. no active seizures, no sedation, haemodynamically stable, etc.)

Exclusion Criteria: Patients who do not meet inclusion criteria above.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Western Neurosensory Stimulation Profile - to assess change in alertness and cognitive functioning | To be administered pre intervention (once consent obtained and prior to intervention - to obtain baseline data) and post intervention (after 4 week intervention period to determine change in alertness/cognitive functioning post intervention).

SECONDARY OUTCOMES:
Ranchos Los Amigos Levels of Cognitive Functioning Scale | To be administered pre intervention (once consent obtained and prior to intervention - to obtain baseline data) and post intervention (after 4 week intervention period to determine change in alertness/cognitive functioning post intervention).
Glasgow Coma Scale | To be administered pre intervention (once consent obtained and prior to intervention - to obtain baseline data) and post intervention (after 4 week intervention period to determine change in alertness/responsiveness post intervention).
Enrollment rates | To be collected during the patient enrollment process (study duration approximately 1 year).
Barriers to enrollment | To be collected during the patient enrollment process (study duration approximately 1 year).
Duration of each intervention session (minutes) | To be collected at the end each intervention session throughout the 4 week intervention period.
Pre/post-intervention heart rate (beats/minute) | To be collected at the beginning and end of each intervention session throughout the 4 week intervention period.
Sp02 reading (percentage) | To be collected at the beginning and end of each intervention session throughout the 4 week intervention period.
Respiratory Rate (breaths/minute) | To be collected at the beginning and end of each intervention session throughout the 4 week intervention period.
ICU Mobility Scale Score | Daily scores are recorded and eventually averaged over 4 week intervention period.
Number of intervention sessions (control or multisensory stimulation) per patient over 4 week period | To be collected at the end of 4 week intervention period.
Barriers to intervention | To be collected (as applicable) at the end of each intervention session throughout the 4 week intervention period.
Date of patient transfer from TNICU to ward | To be collected when patient transferred from TNICU to ward (which may be at any time throughout study period, up to 6 months after study enrollment).
Patient length of stay (days) | To be collected when patient is discharged/transferred from hospital. (which will be at any time, up to 6 months after study enrollment).
Discharge Destination | To be recorded when patient is discharged/transferred from hospital (which will be at any time, up to 6 months after study enrollment).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A St. Louis, BSc, MHSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No